CLINICAL TRIAL: NCT05942079
Title: The Effect of Reiki on Treatment Compliance, Eating Behaviors and Metabolic Values in Obese Individuals With Type 2 Diabetes": Randomized Controlled Study
Brief Title: "The Effect of Reiki on Metabolic Parameters in Obese Type 2 Diabetes Patients''
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Fatmaz zehra KÜÇÜK, PHD STUDENT, Hasan Kalyoncu University
Other Study IDs: 2022/076
Record Dates: First submitted 2023-06-26; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus Type 2 in Obese
Keywords: Reiki; Type 2 DM; Obesity; Eating Behavior; TREATMENT COMPLIANCE BEHAVIORS; NURSING CARE
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group receiving reiki: Individuals who will undergo Reiki for 12 weeks
  Interventions: Other: REİKİ
- control group: control group

INTERVENTIONS:
Other: REİKİ — Reiki is applied as an alternative and complementary treatment method.
  Groups: group receiving reiki

SUMMARY:
The increase in the prevalence of diabetes and the loss of various organs and functions in the individual as a result of complications caused by diabetes affect the life expectancy and quality of individuals, and cause social and economic losses affecting the whole society. For this reason, the individual management of the diabetic patient is important in terms of ensuring effective participation and compliance in treatment and care. Patients must have knowledge, skills and positive attitudes in order to successfully comply with diabetes treatment. Patients are in compliance with diabetes treatment; they encounter some barriers such as medication barriers, barriers to self-monitoring, knowledge and belief barriers, barriers to diagnosis, barriers in relations with health professionals, barriers to lifestyle change, barriers to coping with diabetes, and barriers to getting advice and support. The American Diabetes Association (ADA) states that self-monitoring of blood sugar is important in ensuring glycemic control and preventing hyperglycemia and asymptomatic hypoglycemia. Reiki is applied as an alternative and complementary treatment method. Reiki application, when used together with pharmacological methods, chronic fatigue, diabetic neuropathy, pain caused by surgery, cancer treatment, symptoms of cardiovascular diseases, emotional disorders such as anxiety, depression, acute or chronic pain, infertility-related problems, neurodegenerative disorders, AIDS, autism and developmental disorders, Crohn's disease, irritable bowel syndrome, traumatic brain injury and has been shown to improve health problems such as fatigue.

In the literature, the effects of reiki have been examined in patient groups with different chronic diseases, but no study has been found on obese individuals with Type 2 diabetes. Therefore, reikinin in obese individuals with Type 2 diabetes; This study is planned to determine whether it has an effect on compliance with diabetes treatment, eating behaviors, anxiety levels and changes in metabolic values.

DETAILED DESCRIPTION:
The increase in the prevalence of diabetes and the loss of various organs and functions in the individual as a result of complications caused by diabetes affect the life expectancy and quality of individuals, and cause social and economic losses affecting the whole society. Diabetes with poor management causes many acute and chronic complications. Keeping diabetes under control seriously affects the occurrence of microvascular and macrovascular complications, which develop over years and seriously affect life. Compliance with diabetes treatment; nutrition therapy, regular exercise program, patient self-monitoring, medication, access to health facilities and patient education. With regular monitoring and monitoring of these parameters, compliance with a successful diabetes treatment is improved. The basis of compliance with diabetes treatment is determined by the attitudes and behaviors of patients regarding their own health. For this reason, the individual management of the diabetic patient is important in terms of ensuring effective participation and compliance in treatment and care. Patients must have knowledge, skills and positive attitudes in order to successfully comply with diabetes treatment. Patients are in compliance with diabetes treatment; they encounter some barriers such as medication barriers, barriers to self-monitoring, knowledge and belief barriers, barriers to diagnosis, barriers in relations with health professionals, barriers to lifestyle change, barriers to coping with diabetes, and barriers to getting advice and support. The inability of the individual to cope with these obstacles adequately causes problems in compliance with diabetes treatment. One of the most important points in compliance with diabetes management and treatment is self-monitoring of blood glucose. The American Diabetes Association (ADA) states that self-monitoring of blood sugar is important in ensuring glycemic control and preventing hyperglycemia and asymptomatic hypoglycemia. HbA1c levels were found to be lower in patients who measured their blood glucose more frequently. In patients with poor diabetes management and persistent hyperglycemia, there is an increase in HbA1c value. A 1% increase in HbA1c value is accepted as a risk in the formation of complications. Reiki is applied as an alternative and complementary treatment method. Reiki application, when used together with pharmacological methods, chronic fatigue, diabetic neuropathy, pain caused by surgery, cancer treatment, symptoms of cardiovascular diseases, emotional disorders such as anxiety, depression, acute or chronic pain, infertility-related problems, neurodegenerative disorders, AIDS, autism and developmental disorders, Crohn's disease, irritable bowel syndrome, traumatic brain injury and has been shown to improve health problems such as fatigue (43).

In the literature, the effects of reiki have been examined in patient groups with different chronic diseases, but no study has been found on obese individuals with Type 2 diabetes. Therefore, reikinin in obese individuals with Type 2 diabetes; This study is planned to determine whether it has an effect on compliance with diabetes treatment, eating behaviors, anxiety levels and changes in metabolic values.

ELIGIBILITY:
Inclusion Criteria:

1. Having been diagnosed with Type 2 diabetes at least 6 months ago,
2. Body mass index ≥ 30 kg/m²
3. Being on oral therapy or using insulin,
4. Ability to communicate and read,
5. Volunteering to participate in research

Exclusion Criteria:

1. Not complying with the principle of voluntarism
2. Answering data collection forms incompletely
3. Desire to leave the study at any stage of the study

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Having been diagnosed with Type 2 diabetes at least 6 months ago, Body mass index ≥ 30 kg/m², Being on oral therapy or using insulin
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
"Reiki has a positive effect on adherence to treatment, eating behaviors and metabolic values in obese individuals with type 2 diabetes. | 12 weeks
  Metabolic changes in the patient before and after reiki
Blood glucose level | 12 weeks
  HbA1c change in the patient before and after reiki
Blood cholesterol level | 12 weeks
  Blood cholesterol exchange level
Blood pressure | 12 weeks
  Blood pressure status
Body mass index | 12 weeks
  Body mass index change
Belly circumference measurement | 12 weeks
  waist circumference will be measured with a tape measure
Anxiety level change | 12 weeks
  TO BE EVALUATED BY SCALE
Change in eating behavior | 12 weeks
  The change in eating behavior will be evaluated with a scale
Change in adherence to treatment | 12 weeks
  change in adherence to treatment will be evaluated with a scale

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Harran unv., Sanliurfa
  - Harran Unv, Sanliurfa

IPD SHARING:
Plan to Share IPD: Yes